CLINICAL TRIAL: NCT04940624
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy, Safety, and Tolerability of Soticlestat as Adjunctive Therapy in Pediatric and Young Adult Subjects With Dravet Syndrome (DS)
Brief Title: A Study of Soticlestat as an Add-on Therapy in Children and Young Adults With Dravet Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-935-3001; jRCT2051210074 (Registry Identifier: jRCT); 2021-002480-22 (EudraCT Number)
Record Dates: First submitted 2021-06-16; First posted 2021-06-25 (Actual); Results first posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Dravet Syndrome (DS)
Keywords: Drug Therapy
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — soticlestat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Soticlestat placebo-matching mini-tablets or tablets, orally or via gastrostomy tube (G-tube) or low-profile gastric tube (MIC-KEY) button or jejunostomy tube (J-tube), twice daily (BID), up to 4 weeks during titration. Participants continued to receive the soticlestat placebo-matching mini-tablets or tablets for 12 weeks during maintenance. The total duration of the treatment was up to 16 weeks (Full Treatment Period). Soticlestat matching tapering was done to maintain the blind if participants decided to discontinue the treatment.
  Interventions: Drug: Placebo
- Soticlestat (Experimental): Participants weighing <45 kg: Soticlestat, mini-tablets, at the dose of 40 mg to 200 mg, orally or via G-tube or MIC-KEY button or J-tube, BID based on the body weight up to 4 weeks during titration. Participants continued to receive the dose that they were on at the end of the titration, for 12 weeks during maintenance. The total duration of the treatment was up to 16 weeks (Full Treatment Period) with dose tapered down if participants decided to discontinue the treatment.
  Participants weighing ≥45 kg: Soticlestat mini-tablets or tablets with a starting dose of 100 mg BID followed by 200 mg BID and, then 300 mg BID, up to 4 weeks during titration. Participants continued to receive 300 mg BID for 12 weeks during maintenance. The total duration of the treatment was up to 16 weeks (Full Treatment Period) with dose tapered down if participants decided to discontinue the treatment.
  Interventions: Drug: Soticlestat

INTERVENTIONS:
Drug: Soticlestat — Soticlestat mini-tablets or tablets.
  Other Names: TAK-935
  Arms: Soticlestat
Drug: Placebo — Soticlestat placebo-matching mini-tablets or tablets.
  Arms: Placebo

SUMMARY:
The main aim of the study is to learn if soticlestat, when given as an add-on therapy, reduces the number of convulsive seizures in children and young adults with DS.

Participants will receive their standard antiseizure therapy, plus either a tablet of soticlestat or placebo for 16 weeks. A placebo looks just like soticlestat but will not have any medicine in it.

Participants may continue treatment in an extension study, based on the extension study's entry criteria. Those that want to stop treatment will have a gradual dose reduction during 1 week and then be followed up for 2 weeks.

DETAILED DESCRIPTION:
The drug being tested in this study is called soticlestat (TAK-935). Soticlestat as an adjunctive therapy will be assessed for efficacy, safety, and tolerability in pediatric and adult participants with DS.

The study will enroll approximately 142 pediatric and young adult patients. Participants will be randomized at a 1:1 ratio to receive standard of care (SOC) plus one of the following adjunctive therapies:

* Soticlestat or
* Placebo

The total daily dose of study drug will be calculated based on body weight in the 4 weeks Titration Period. Following the Titration Period, participants will continue to receive the same dose in the 12-weeks Maintenance Period.

This multi-center trial will be conducted worldwide. The overall time to participate in the study will be from 22-25 weeks. At the end of the Full Treatment Period, participants have the option to either complete the study and taper off the investigational product or to enter the OLE if they meet eligibility requirements. If participants discontinue, they will be followed-up on phone call approximately 14 days after the last dose of study drug for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Has documented clinical diagnosis of DS.
2. Had ≥12 convulsive seizures over 12 weeks before screening based on the historical information and has had ≥4 convulsive seizures per 28 days during the 4- to 6-week prospective baseline period.
3. Weighs ≥10 kg at the screening visit (Visit 1).
4. Failure to control seizures despite appropriate trials of at least 1 ASM based on historical information and is currently on an antiseizure therapy or other treatment options considered as SOC.
5. Artisanal cannabidiols are allowed at a stable dose for at least 4 weeks before the screening visit (Visit 1); the dosing regimen and manufacturer should remain constant throughout the study (Artisanal cannabidiols will not be counted as ASMs.).
6. Currently taking 0 to 4 ASMs at stable doses for at least 4 weeks before the screening visit (Visit 1); benzodiazepines used chronically (daily) to treat seizures are considered ASMs. Fenfluramine and cannabidiol (Epidiolex) are allowed where available and should be counted as an ASM. ASM dosing regimen must remain constant throughout the study.

Exclusion Criteria:

1. Unstable, clinically significant neurologic (other than the disease being studied), psychiatric, cardiovascular, ophthalmologic, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, hematopoietic, endocrine disease, malignancy including progressive tumors, or other abnormality that may impact the ability to participate in the study or that may potentially confound the study results. It is the responsibility of the investigator to assess the clinical significance; however, consultation with the medical monitor may be warranted.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (66):
- United States (10):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California Benioff Children's Hospital, San Francisco, California
  - Clinical Integrative Research Center of Atlanta, Atlanta, Georgia
  - University of Iowa Hospitals & Clinics - (CRS), Iowa City, Iowa
  - NYU Comprehensive Epilepsy Center, New York, New York
  - University of Toledo, Toledo, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Seattle Children's Hospital, Seattle, Washington
  - Multicare Health System - Mary Bridge Pediatrics, Tacoma, Washington
- Queensland Childrens Hospital, South Brisbane, Queensland, Australia
- Brazil (3):
  - Instituto de Neurologia de Curitiba (INC), Curitiba, Paraná
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre, Rio Grande do Sul
  - Universidade de Sao Paulo, São Paulo
- Canada (3):
  - Alberta Childrens Hospital, Calgary, Alberta
  - Child and Family Research Institute, Vancouver, British Columbia
  - Hospital For Sick Children, Toronto, Ontario
- China (10):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Children's Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Wuhan Childrens hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Hospital of Jilin University, Changchun, Jilin
  - Children's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
- France (3):
  - Hopitaux de La Timone, Marseille
  - Hopital Necker - Enfants Malades, Paris
  - Hopital Robert Debre, Paris
- Germany (3):
  - Schon Klinik Vogtareuth, Vogtareuth, Bavaria
  - Klinikum der Johann-Wolfgang Goethe-Universitat, Frankfurt am Main, Hesse
  - Krankenhaus Mara gGmbH - Epilepsiezentrum Bethel, Bielefeld, North Rhine-Westphalia
- Attikon University General Hospital, Chaïdári, Attica, Greece
- Orszagos Mentalis, Ideggyogyaszati es Idegsebeszeti Intezet, Budapest, Hungary
- Italy (4):
  - IRCCS Ospedale Pediatrico Bambino Gesu - INCIPIT - PIN, Rome, Lazio
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - ASST di Pavia - Fondazione Istituto Neurologico Mondino IRCCS, Pavia, Lombardy
  - Azienda Ospedaliero Universitaria A Meyer - INCIPIT - PIN, Florence, Tuscany
- Japan (9):
  - Aichi Medical University Hospital, Nagakute-Shi, Aiti
  - Kumamoto-Ezuko Medical Center for The Severely Disabled, Kumamoto, Kumamoto
  - National Hospital Organization Nagasaki Medical Center, Omura-Shi, Nagasaki
  - National Hospital Organization Nishi-Niigata Chuo National Hospital, Niigata, Niigata
  - Osaka City General Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita-Shi, Osaka
  - National Hospital Organization Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka, Shizuoka
  - Hokkaido University Hospital, Chuo-Ku, Tokyo
  - National Center of Neurology and Psychiatry, Kodaira-Shi, Tokyo
- Childrens University Hospital, Riga, Latvia
- Netherlands (2):
  - Kempenhaeghe - PPDS, Heeze, North Brabant
  - Stichting Epilepsie Instellingen Nederland, Zwolle, Overijssel
- Poland (4):
  - Centrum Medyczne Plejady, Krakow, Lesser Poland Voivodeship
  - Neurosphera SP. Z O.O, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpital Kliniczny im. H.Swiecickiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
- Russia (2):
  - Russian National Research Medical University n.a. N.I.Pirogov, Moscow, Moscow
  - Krasnoyarsk State Medical University n.a. V.F. Voyno-Ysenetskiy, Krasnoyarsk
- Serbia (3):
  - Clinic for Neurology and Psychiatry for Children and Youth, Belgrade
  - Mother and Child Health Care Institute of Serbia Dr Vukan Cupic, Belgrade
  - University Clinical Center Nis, Niš
- Spain (3):
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Regional Universitario de Malaga Hospital General, Málaga
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Ukraine (3):
  - Communal Non-profit Enterprise City Childrens Clinical Hospital #6 of DCC, Dnipro, Dnipropetrovsk Oblast
  - Communal Non-commercial Enterprise Iv-Frank Regional Childrens Clinical Hosp of Iv-Frank RC, Ivano-Frankivsk
  - CNPE Clinical Hospital Psychiatry of the Executive Body of the Kyiv City Council KCSA, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60e40858ef0b71001e743e10

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 144 participants participated in the study at multiple investigative sites globally from 28 October 2021 to 11 April 2024.
Pre-assignment Details: A total of 144 participants with a diagnosis of Dravet Syndrome (DS) were randomized in a 1:1 ratio to receive either soticlestat or placebo.
Period: Overall Study
Arm/Group | Placebo | Soticlestat
Started | 71 | 73
Completed | 63 | 60
Not Completed | 8 | 13
Not completed — Adverse Event | 4 | 11
Not completed — Withdrawal by Parent/Guardian | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Reason Not Specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who had taken at least one dose of study drug.
Groups:
- Placebo: Soticlestat placebo-matching mini-tablets or tablets, orally or via G-tube or MIC-KEY button or J-tube, BID, up to 4 weeks during titration. Participants continued to receive the soticlestat placebo-matching mini-tablets or tablets for 12 weeks during maintenance. The total duration of the treatment was up to 16 weeks (Full Treatment Period). Soticlestat matching tapering was done to maintain the blind if participants decided to discontinue the treatment.
- Total: Total of all reporting groups
Arm/Group | Placebo | Soticlestat | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (5.06) | 10.1 (5.04) | 10.3 (5.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 36 | 36 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 62 | 68 | 130
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 24 | 27 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 43 | 39 | 82
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Convulsive Seizure Frequency Per 28 Days During the Full Treatment Period
Description: Convulsive seizure frequency per 28 days was defined as the total number of convulsive seizures reported during the period divided by the number of days during the period seizures were assessed multiplied by 28. Percent change from Baseline was defined as (frequency of seizures per 28 days during the Full Treatment Period - frequency of seizures per 28 days at Baseline) divided by the frequency of seizures per 28 days at Baseline multiplied by 100.
Time Frame: Baseline; Full Treatment Period: Weeks 1 to 16
Population: Modified Intent-to-Treat (mITT) Analysis Set included all randomized participants who had received at least one dose of study drug and had been assessed for seizures for at least one day in the Full Treatment Period.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 71 | 73
percent change | -8.64 [-30.13 to 14.83] | -22.16 [-53.64 to 22.73]
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; p = 0.061, ANCOVA — The p-value was calculated by Rank Analysis of Covariance (ANCOVA) model using treatment group, age stratum (≤6 years, >6 years), and rank of Baseline seizure frequency per 28 days as predictors; Hodges-Lehmann Location Shift Estimate = -15.64, 95% CI 2-sided [-31.30 to 0.24] — The location shift between soticlestat and placebo (soticlestat - placebo) and its asymptotic 95% confidence interval (CI) were based on the Hodges-Lehmann estimation

2. Primary Outcome: Percent Change From Baseline in Convulsive Seizure Frequency Per 28 Days During the Maintenance Period
Description: Convulsive seizure frequency per 28 days was defined as the total number of convulsive seizures reported during the period divided by number of days during the period seizures were assessed multiplied by 28. Percent change from Baseline was defined as (frequency of seizures per 28 days during Maintenance Period - frequency of seizures per 28 days at Baseline) divided by the frequency of seizures per 28 days at Baseline multiplied by 100.
Time Frame: Baseline; Maintenance Period: Weeks 5 to 16
Population: mITT Analysis Set included all randomized participants who had received at least one dose of study drug and had been assessed for seizures for at least one day in the Full Treatment Period. Overall number of participants analyzed indicates the number of participants with data available for analyses.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 68 | 69
percent change | -11.99 [-31.93 to 9.75] | -23.29 [-56.92 to 14.15]
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; p = 0.089, ANCOVA — The p-value was calculated by the Rank ANCOVA model using treatment group, age stratum (≤6 years, >6 years), and rank of baseline seizure frequency per 28 days as predictors; Hodges-Lehmann Location Shift Estimate = -14.29, 95% CI 2-sided [-30.51 to 1.53] — The location shift between soticlestat and placebo (soticlestat - placebo) and its asymptotic 95% CI were based on the Hodges-Lehmann estimation

3. Secondary Outcome: Percentage of Responders During Maintenance Period
Description: Responders were defined as those with ≥50% reduction from Baseline in convulsive seizures during the Maintenance Period. Percentages were rounded off to the nearest single decimal place.
Time Frame: Maintenance Period: Weeks 5 to 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 68 | 69
percentage of participants | 11.8 | 30.4
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; p = 0.010, Cochran-Mantel-Haenszel; The p-value was based on Cochran-Mantel-Haenszel (CMH) test stratified by age stratum (≤6 years, >6 years); Odds Ratio (OR) = 3.22, 95% CI 2-sided [1.30 to 7.96]

4. Secondary Outcome: Percentage of Responders During the Full Treatment Period
Description: Responders were defined as those with ≥50% reduction from Baseline in convulsive seizures during the Full Treatment Period. Percentages were rounded off to the nearest single decimal place.
Time Frame: Full Treatment Period: Weeks 1 to 16
Population: mITT Analysis Set included all randomized participants who had received at least one dose of study drug and had been assessed for seizures for at least one day in the Full Treatment Period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 71 | 73
percentage of participants | 9.9 | 27.4
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; p = 0.008, Cochran-Mantel-Haenszel; The p-value was based on CMH test stratified by age stratum (≤6 years, >6 years); Odds Ratio (OR) = 3.59, 95% CI 2-sided [1.36 to 9.49]

5. Secondary Outcome: Percentage of Participants With ≤0%, >0% to ≤25%, >25% to ≤50%, >50% to ≤75%, and >75% to ≤100% Reduction in Convulsive Seizures During the Full Treatment Period
Description: Percent reduction from Baseline (%) was defined as [(Full Treatment Period Convulsive Seizure Frequency - Baseline Convulsive Seizure Frequency) divided by Baseline Convulsive Seizure Frequency] multiplied by 100. Data was reported as reduction of ≤0%, >0% to ≤25%, >25% to ≤50%, >50% to ≤75%, >75% to ≤100% or more in seizures from Baseline. Percentages were rounded off to the nearest single decimal place.
Time Frame: Full Treatment Period: Weeks 1 to 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 71 | 73
percentage of participants
  ≤0% Reduction | 39.4 | 31.5
  >0% to ≤25% Reduction | 32.4 | 20.5
  >25% to ≤50% Reduction | 18.3 | 20.5
  >50% to ≤75% Reduction | 8.5 | 13.7
  >75% to ≤100% Reduction | 1.4 | 13.7

6. Secondary Outcome: Percentage of Participants With Caregiver Global Impression of Improvement (Care GI-I) Scale Responses as Per the Parent/Caregiver Reported Impression at Week 16
Description: The Care GI-I is a 7-point Likert scale that the caregiver used to rate improvement in overall seizure control, behavior, safety and tolerability after the initiation of study drug relative to Baseline (before treatment with the study drug). The participant was rated as follows: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), and 7 (very much worse). The parent/caregiver completed the Care GI-I via interview. Lower scores indicate improvement. Percentages were rounded off to the nearest single decimal place.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 68 | 66
percentage of participants
  Score 1: Very Much Improved | 1.5 | 4.5
  Score 2: Much Improved | 11.8 | 27.3
  Score 3: Minimally Improved | 22.1 | 28.8
  Score 4: No Change | 47.1 | 27.3
  Score 5: Minimally Worse | 10.3 | 7.6
  Score 6: Much Worse | 5.9 | 3.0
  Score 7: Very Much Worse | 1.5 | 1.5
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; p = 0.004, Cumulative Logit Model; P-value was calculated using the Cumulative Logit model including treatment and age group as factors; Odds Ratio (OR) = 2.51, 95% CI 2-sided [1.33 to 4.72]

7. Secondary Outcome: Percentage of Participants With Clinical Global Impression of Improvement (CGI-I) Scale Responses as Per the Investigator Reported Impression at Week 16
Description: The CGI-I (Clinician) is a 7-point Likert scale that the investigator used to rate a participant's change (improvement) in overall seizure control, behavior, safety and tolerability, after the initiation of study drug relative to Baseline (before treatment with the study drug). The participant was rated as follows: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), and 7 (very much worse). The investigator or designee completed the CGI-I. Lower scores indicate improvement. Percentages were rounded off to the nearest single decimal place.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 71 | 71
percentage of participants
  Score 1: Very Much Improved | 2.8 | 7.0
  Score 2: Much Improved | 8.5 | 25.4
  Score 3: Minimally Improved | 15.5 | 19.7
  Score 4: No Change | 59.2 | 38.0
  Score 5: Minimally Worse | 5.6 | 8.5
  Score 6: Much Worse | 8.5 | 1.4
  Score 7: Very Much Worse | 0.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; p = 0.003, Cumulative Logit Model; P-value was calculated using the Cumulative Logit model including treatment and age group as factors; Odds Ratio (OR) = 2.58, 95% CI 2-sided [1.37 to 4.87]

8. Secondary Outcome: Percentage of Participants With CGI-I Nonseizure Symptoms Instrument Responses for Each Domain as Per the Investigator Reported Impression at Week 16
Description: The CGI-I non-seizure symptoms instrument is a series of single-item assessments that the investigator used to rate improvement in the symptoms and impacts in select non-seizure domains (alertness, communication, and disruptive behaviors) since initiating the study drug. The participant was rated by the investigator for each domain as follows: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), and 7 (very much worse). Lower scores indicated improvement. Data for percentage of participants categorized based on the responses for each domain are presented. Percentages were rounded off to the nearest single decimal place.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 71 | 71
percentage of participants
  Alertness: Score 1: Very Much Improved | 2.8 | 7.0
  Alertness: Score 2: Much Improved | 8.5 | 4.2
  Alertness: Score 3: Minimally Improved | 14.1 | 14.1
  Alertness: Score 4: No Change | 67.6 | 70.4
  Alertness: Score 5: Minimally Worse | 5.6 | 4.2
  Alertness: Score 6: Much Worse | 1.4 | 0.0
  Alertness: Score 7: Very Much Worse | 0.0 | 0.0
  Communication: Score 1: Very much Improved | 1.4 | 4.2
  Communication: Score 2: Much Improved | 11.3 | 5.6
  Communication: Score 3: Minimally Improved | 18.3 | 22.5
  Communication: Score 4: No Change | 62.0 | 62.0
  Communication: Score 5: Minimally Worse | 4.2 | 4.2
  Communication: Score 6: Much Worse | 2.8 | 1.4
  Communication: Score 7: Very Much Worse | 0.0 | 0.0
  Disruptive Behaviors: Score 1: Very Much Improved | 1.4 | 1.4
  Disruptive Behaviors: Score 2: Much Improved | 4.2 | 5.6
  Disruptive Behaviors: Score 3: Minimally Improved | 14.1 | 16.9
  Disruptive Behaviors: Score 4: No Change | 69.0 | 64.8
  Disruptive Behaviors: Score 5: Minimally Worse | 11.3 | 8.5
  Disruptive Behaviors: Score 6: Much Worse | 0.0 | 1.4
  Disruptive Behaviors: Score 7: Very Much Worse | 0.0 | 1.4
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Alertness; Test type: Superiority; p = 0.741, Cumulative Logit Model; P-value was calculated using the Cumulative Logit model including treatment and age group as factors; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.56 to 2.26]
Statistical Analysis 2: Comparison: Placebo vs Soticlestat; Communication; Test type: Superiority; p = 0.901, Cumulative Logit Model; P-value was calculated using the Cumulative Logit model including treatment and age group as factors; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.54 to 2.02]
Statistical Analysis 3: Comparison: Placebo vs Soticlestat; Disruptive Behaviors; Test type: Superiority; p = 0.693, Cumulative Logit Model; P-value was calculated using the Cumulative Logit model including treatment and age group as factors; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.58 to 2.28]

9. Secondary Outcome: Change From Baseline in Quality of Life Inventory-Disability (QI-Disability) Total Score at Week 16
Description: The QI-Disability tool is a parent/caregiver-reported questionnaire that evaluated the quality of life in children with intellectual disabilities. It contains 32 items covering 6 domains of quality of life: physical health, positive emotions, negative emotions, social interaction, leisure and the outdoors, and independence. Each QI-Disability item is rated on a Likert scale of: Never, Rarely, Sometimes, Often, and Very Often. Items were linearly transformed to a scale of 0 to 100, with higher scores representing better quality of life. Domain scores are calculated by averaging item scores. The domain scores are summed and divided by 6 to yield a total score. The total score ranges from 0 to 100, with higher scores indicating a better quality of life. A negative change from Baseline implies deteriorating quality of life. Mixed-effects model for repeated measures (MMRM) was used for analysis.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 53 | 56
score on a scale | 2.81 (10.119) | -1.23 (15.438)
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; p = 0.189, MMRM — P-value was based on MMRM analysis with change from baseline as outcome and baseline score as fixed continuous effect; treatment group, age stratum, analysis visit, and analysis visit by treatment group interaction as fixed categorical effects; Least Square Mean Difference = -3.03, 95% CI 2-sided [-7.59 to 1.52]

10. Secondary Outcome: Percentage of Participants With CGI-I Seizure Intensity and Duration Instrument Responses as Per the Parent/Caregiver Reported Impression at Week 16
Description: The CGI-I seizure intensity and duration instrument was used by the parent/caregiver to rate changes in intensity and/or duration of the most impactful seizures from the first assessment. The participant's symptoms were rated on 7-point scale as follows: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), and 7 (very much worse). Lower scores indicate improvement. Percentages were rounded off to the nearest single decimal place.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 69 | 65
percentage of participants
  Score 1: Very Much Improved | 4.3 | 10.8
  Score 2: Much Improved | 4.3 | 24.6
  Score 3: Minimally Improved | 15.9 | 23.1
  Score 4: No Change | 59.4 | 33.8
  Score 5: Minimally Worse | 5.8 | 1.5
  Score 6: Much Worse | 8.7 | 6.2
  Score 7: Very Much Worse | 1.4 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; p < 0.001, Cumulative Logit Model; P-value was calculated using the Cumulative Logit model including treatment and age group as factors; Odds Ratio (OR) = 3.65, 95% CI 2-sided [1.87 to 7.13]

11. Secondary Outcome: Percent Change From Baseline in Frequency of All Seizures Per 28 Days During the Maintenance Period
Description: Seizure frequency per 28 days was defined as the total number of seizures reported during the period divided by the number of days during the period seizures were assessed multiplied by 28. Percent change from Baseline was defined as (frequency of seizures per 28 days during the Maintenance Period - frequency of seizures per 28 days at Baseline) divided by the frequency of seizures per 28 days at Baseline multiplied by 100.
Time Frame: Baseline; Maintenance Period: Weeks 5 to 16
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 68 | 69
percent change | -11.89 [-33.78 to 10.50] | -17.24 [-56.83 to 23.70]
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; p = 0.565, ANCOVA; The Rank ANCOVA model used treatment group, age stratum (≤6 years, >6 years), and rank of Baseline seizure frequency per 28 days as predictors; Hodges-Lehmann Location Shift Estimate = -9.97, 95% CI 2-sided [-29.01 to 7.87] — [estimate comment as in outcome 2, analysis 1]

12. Secondary Outcome: Percent Change From Baseline in Frequency of All Seizures Per 28 Days During the Full Treatment Period
Description: Seizure frequency per 28 days was defined as the total number of seizures reported during the period divided by number of days during the period seizures were assessed multiplied by 28. Percent change from Baseline was defined as (frequency of seizures per 28 days during the Full Treatment Period - frequency of seizures per 28 days at Baseline) divided by the frequency of seizures per 28 days at Baseline multiplied by 100.
Time Frame: Baseline; Full Treatment Period: Weeks 1 to 16
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 71 | 73
percent change | -7.46 [-32.37 to 14.83] | -9.27 [-54.11 to 30.00]
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; p = 0.637, ANCOVA; [statistical method as in outcome 11, analysis 1]; Hodges-Lehmann Location Shift Estimate = -8.13, 94% CI 2-sided [-26.31 to 10.13] — [estimate comment as in outcome 2, analysis 1]

13. Secondary Outcome: Change From Baseline in Percentage of Convulsive Seizure-free Days During the Full Treatment Period
Description: Convulsive seizure-free days was defined as number of days a participant remained convulsive seizure-free after initiation of the treatment. The change from baseline in percentage of convulsive seizure-free days, was defined as the percentage of seizure-free days during the Full Treatment Period minus the percentage of seizure-free days during the Baseline. A linear model with treatment group and age stratum as factors and baseline percentage as a covariate was used for analysis.
Time Frame: Baseline up to Week 16
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 71 | 73
percentage of days | 2.74 (1.784) | 3.54 (1.719)
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; Least Square Mean Difference = 0.79, 95% CI 2-sided [-3.81 to 5.40] — A linear model with treatment group and age stratum as factors and baseline percentage as a covariate was used for analysis

14. Secondary Outcome: Longest Convulsive Seizure-free Interval During the Full Treatment Period
Description: Longest convulsive seizure-free interval was defined as the longest time period that the participant remained convulsive seizure free after initiation of the treatment. A linear model with treatment group and age stratum as factors was used for analysis.
Time Frame: Full Treatment Period: Weeks 1 to 16
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 71 | 73
days | 16.7 (2.15) | 22.3 (2.08)
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; Least Square Mean Difference = 5.6, 95% CI 2-sided [0.1 to 11.2]

15. Secondary Outcome: Number of Days When Rescue Antiseizure Medication (ASM) is Used During the Full Treatment Period
Description: Use of rescue ASM was recorded in the case report form (CRF) along with start and end date of medication. Based on the start and end dates for all rescue ASMs taken by a participant, the number of days during the Full Treatment Period when rescue ASM was used was derived.
Time Frame: Full Treatment Period: Weeks 1 to 16
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 71 | 73
days | 4.0 (0.81) | 2.9 (0.78)
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; Least Square Mean Difference = -1.1, 95% CI 2-sided [-3.1 to 1.0] — Least square mean difference was estimated using a linear model with treatment group and age stratum as factors

ADVERSE EVENTS:
Time Frame: From the first dose up to Week 19
Description: Safety Analysis Set included all participants who had taken at least one dose of study drug.
Arm/Group | Placebo | Soticlestat
All-Cause Mortality (participants affected / at risk) | 0/71 | 1/73
Serious Adverse Events (participants affected / at risk) | 10/71 | 7/73
Other Adverse Events (participants affected / at risk) | 37/71 | 40/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | Soticlestat (N=73)
Adenovirus infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Seizure (Nervous system disorders) | 1 | 0
Seizure cluster (Nervous system disorders) | 1 | 2
Status epilepticus (Nervous system disorders) | 4 | 2
Sudden unexplained death in epilepsy (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | Soticlestat (N=73)
Change in seizure presentation (Nervous system disorders) | 9 | 10
Constipation (Gastrointestinal disorders) | 0 | 6
Decreased appetite (Metabolism and nutrition disorders) | 4 | 5
Fatigue (General disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 1 | 6
Nasopharyngitis (Infections and infestations) | 9 | 9
Pyrexia (General disorders) | 9 | 8
Somnolence (Nervous system disorders) | 8 | 10
Upper respiratory tract infection (Infections and infestations) | 8 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT04940624/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT04940624/SAP_001.pdf